CLINICAL TRIAL: NCT00876616
Title: An Multi-site, Open, Prospective Study to Assess the Efficacy and Safety of Multi-target Therapy in the Treatment of Class Ⅲ,Ⅳ,Ⅴ,Ⅲ+Ⅴand Ⅳ+Ⅴ Lupus Nephritis
Brief Title: Assess the Efficacy and Safety of Multi-target Therapy in Lupus Nephritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhi-Hong Liu, M.D. (Other)
Collaborators: Ruijin Hospital (Other); West China Hospital (Other); RenJi Hospital (Other); China Medical University, China (Other); Huashan Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Beijing Friendship Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Zhi-Hong Liu, M.D., professor, Nanjing University School of Medicine
Organization: Nanjing University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0901
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Lupus Nephritis
Keywords: lupus nephritis;multi-target therapy; MMF; FK506
MeSH Terms: conditions — Lupus Nephritis | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus+Mycophenolate mofetil (Experimental): FK506 4mg/d+MMF 1.0g/d
  Interventions: Drug: Tacrolimus+Mycophenolate mofetil
- Cyclophosphamide (Active Comparator): CTX iv 0.75 g/m2 body surface area (BSA)
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Tacrolimus+Mycophenolate mofetil — FK506 4mg/d,MMF 1.0g/d
  Other Names: FK506+MMF
  Arms: Tacrolimus+Mycophenolate mofetil
Drug: Cyclophosphamide — CTX 0.75g/m2 BSA
  Other Names: CTX
  Arms: Cyclophosphamide

SUMMARY:
The purpose of this study is to assess the efficacy and safety of multi-target therapy in the treatment of class Ⅲ,Ⅳ,Ⅴ,Ⅲ+Ⅴand Ⅳ+Ⅴ lupus nephritis.

DETAILED DESCRIPTION:
1. To assess the efficacy of FK506 combined with MMF vs intravenous cyclophosphamide (CTX) pulses in treatment of class Ⅲ,Ⅳ,Ⅴ,Ⅲ+Ⅴand Ⅳ+Ⅴ Lupus Nephritis (LN).
2. To investigate the safety and tolerability of FK506 combined with MMF vs intravenous CTX pulses in the treatment of class Ⅲ,Ⅳ,Ⅴ,Ⅲ+Ⅴand Ⅳ+Ⅴ LN.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent by subject or guardian
2. 18 to 65 years of age (inclusive 18 and 65), male or female
3. Diagnosis of SLE according to the American College of Rheumatology criteria (1997)
4. Diagnosis of Class Ⅲ,Ⅳ,Ⅴ,Ⅲ+Ⅴand Ⅳ+ⅤLN according to the ISN/RPS 2003 classification by light, immunofluorescence, and electron microscopy within 6 months before enrollment
5. Pathologic chronic index (CI) ≤3' without thrombotic microangiopathy (TMA)
6. SLE Disease Activity Index (DAI) >10'
7. Proteinuria ≥1.5g/d，with or without active urinary sediment
8. Serum creatinine (Scr)≤3.0mg/dl (265.2 mol/L)

Exclusion Criteria:

1. Previous treatment with MMF, CTX, tacrolimus, Cyclosporin A (CsA), large doses of immunoglobulin and methylprednisolone (MP), plasmapheresis or renal replacement therapy within the past 12 weeks. Oral glucocorticoids, azathioprine, intravenous MP (≤80mg/d)， short-time CsA (<2 weeks) or leflunomide (<4 weeks) are allowed
2. ALT or AST increase twice above the upper limit of the normal range
3. Hyperglycemia is defined as fasting blood glucose level ≥7.0 mmol/L and/or postprandial blood sugar level>11.1 mmol/L
4. Known hypersensitivity or contraindication to any components of MMF, tacrolimus, CTX or glucocorticoids
5. History of present illness:

   1. active HBV infection (HBsAg, HBeAg and anti-HBc positive or HBsAg, anti- HBe and anti-HBc positive), HCV infection, pulmonary tuberculosis, cytomegalovirus(CMV) infection (defined as CMV-IgM positive or CMV-DNA positive), fungal infection or HIV infection, within 3 months before the enrollment
   2. non-healed active peptic ulcer within 3 months before the enrollment
   3. drug or drinking abuse
   4. malnutrition (BMI <18.5kg/m2) or body weight <50Kg
6. Other active diseases, such as:

   1. severe cardiovascular diseases
   2. chronic obstructive pulmonary disease(COPD)or asthma requiring oral glucocorticoids
   3. marrow depression not due to SLE activation: white blood cell count <3000/mm3 or neutrophil count <1300/mm3 or platelet count <50000/mm3
7. Severe infection or need of antibiotic therapy
8. Female patients who are pregnant/breastfeeding or those patients (both gender) who refused contraception
9. Life-threatening complications such as large hydropericardium, pneumohemorrhagia, lupus encephalopathy and severe pulmonary hypertension or patients in need of MP pulse (>0.5g/d ) treatment because of aggravation of SLE
10. Known to be non-compliance or violation of the protocol base on investigator's judgement
11. Patient who participate of any other investigational drug study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2009-04; Primary Completion 2011-05 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of FK506 combined with MMF vs intravenous CTX pulses in treatment of class Ⅲ, Ⅳ,Ⅴ, Ⅲ+Ⅴand Ⅳ+Ⅴ LN. | 24 weeks
  The primary endpoint is the rate of complete remission at 24 weeks.

SECONDARY OUTCOMES:
To investigate the other efficacy indicators of FK506 combined with MMF vs intravenous CTX pulses in the treatment of class Ⅲ, Ⅳ,Ⅴ, Ⅲ+Ⅴand Ⅳ+Ⅴ LN. | 24 weeks
  The secondary endpoints include total remission, time to complete remission and remission, rate of complete remission and remission in patients with different types of LN, changes between baseline and after 24 week of induction treatment in proteinuria, albumin, SCr, eGFR, complement, autoantibodies, SLE-DAI and dosage and concentration of immunosuppressants between groups.

OTHER OUTCOMES:
To assess the Safety of FK506 combined with MMF vs intravenous CTX pulses in treatment of class Ⅲ, Ⅳ,Ⅴ, Ⅲ+Ⅴand Ⅳ+Ⅴ LN. | 24 weeks
  Safety assessments include clinical manifestations, physical examination, laboratory tests laboratory tests (including hematology, serum chemistry, urinalysis), adverse events (including gastrointestinal toxicity and severe infections requiring antibiotics treatment) and concomitant medications.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, Master, Principal Investigator — Nanjing University School of Medicine
Locations (1):
- Research Institute of Nephrology,Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Liu Z, Zhang H, Liu Z, Xing C, Fu P, Ni Z, Chen J, Lin H, Liu F, He Y, He Y, Miao L, Chen N, Li Y, Gu Y, Shi W, Hu W, Liu Z, Bao H, Zeng C, Zhou M. Multitarget therapy for induction treatment of lupus nephritis: a randomized trial. Ann Intern Med. 2015 Jan 6;162(1):18-26. doi: 10.7326/M14-1030. PMID 25383558